CLINICAL TRIAL: NCT04328350
Title: Social Experiences of Adolescents and Young Adults With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CONNECT
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Childhood Cancer; Social Behavior; Social Competence
MeSH Terms: conditions — Neoplasms; Social Behavior; Social Skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AYA who are on treatment 2-12 months post -diagnosis: AYA will complete questionnaires assessing peer versus family connectedness, peer/romantic competence, coping, distress, social support, and quality of life.A study-specific needs assessment regarding interest in social functioning interventions will also be completed.
  Participants (30 on-therapy) will be interviewed to further explore aspects of peer/family connectedness and intervention interest.
- AYA who are off -therapy 1 to 4 years: AYA will complete questionnaires assessing peer versus family connectedness, peer/romantic competence, coping, distress, social support, and quality of life.A study-specific needs assessment regarding interest in social functioning interventions will also be completed.
  Participants (20 off-therapy) will be interviewed to further explore aspects of peer/family connectedness and intervention interest.

SUMMARY:
Participants are being asked to take part in this clinical trial, a type of research study, because investigators want to learn more about the social experiences adolescents and young adults who are being treated or have been treated for cancer.

Primary Objectives

* Describe differences in social experience variables (peer connectedness, perceived social competence, parent versus peer attachment) based on treatment status: on versus off therapy.
* In on-therapy patients, describe differences in social experience variables (peer connectedness, perceived social competence, parent versus peer attachment) based on developmental stage: high school versus post-high school.

Secondary Objectives

* Assess the social support and peer interaction needs of AYA with cancer as a means of determining stakeholder interest and need for psychosocial interventions targeting social experiences.
* Using qualitative interviews, explore patient perceptions of the impact of cancer on social experiences among AYA, particularly with regards to changes in friendships as a result of the cancer diagnosis and the role of the hospital in helping or hindering friendship maintenance/development.

Exploratory Objectives

* Explore differences in social experience by demographic, disease and treatment factors, including: gender, diagnostic category (brain tumor, leukemia/lymphoma, solid tumor), late effects/symptom burden, and treatment (e.g., treatment intensity, serious medical events).
* Explore associations between perceived impact of cancer and social experience in AYA.
* Explore associations between use of social media and social experience.
* Explore associations between social experiences and overall functioning (quality of life, distress, coping).
* Explore the possibility of subclasses of AYA by using person-centered analyses to empirically derive profiles of social experience.

DETAILED DESCRIPTION:
A mixed-methods design involving questionnaires and interviews will be used to evaluate the study objectives. AYA ages 15 to 22 will be recruited to participate. Two cohorts will be enrolled: AYA who are on-treatment, 2-12 months post-diagnosis; and AYA who are off-therapy 1 to 4 years. AYA will complete questionnaires assessing peer versus family connectedness, peer/romantic competence, coping, distress, social support, and quality of life. A study-specific needs assessment regarding interest in social functioning interventions will also be completed. If a caregiver is available, they will be asked to complete questionnaires regarding family functioning and quality of life. A subset of 50 AYA (30 on-therapy/20 off-therapy) will be interviewed to further explore aspects of peer/family connectedness and intervention interest. Analyses will focus on describing how aspects of social experiences (peer connectedness, social competence, peer versus parent attachment) differ based on treatment status (on versus off therapy) and developmental stage (high school versus post-high school), as well as potential moderators.

Two cohorts of AYA with cancer, ages 15-22, will be identified and recruited for the study: 1) patients on-therapy, 2-12 months from diagnosis; and 2) patients off- therapy 1-4 years, and ≥13 years of age at diagnosis. AYA from all diagnostic groups - brain tumor, solid tumor, leukemia/lymphoma - and developmental periods - high school, post-high school - will be targeted, and care will be taken to ensure a representative sample.

ELIGIBILITY:
Inclusion Criteria:

* All Participants
* Age 15 - 22
* Primary oncology diagnosis.
* Reads and speaks English.
* On-Therapy Strata

  * 2 - 12 months from diagnosis and receiving cancer-directed therapy.
* Off-Therapy Strata

  * 1 - 4 years post-treatment, diagnosed at ≥13 years of age.
* Caregivers Reads and speaks English
* Consent received from adult participant to contact, as it applies

Exclusion Criteria:

* Surgery only treatment plan.
* IQ less than 70 as documented in the medical record.
* Diagnosis of a genetic disorder/pre-existing neurodevelopmental condition associated with neurocognitive or social impairment (e.g., autism, Neurofibromatosis Type 1 (NF1), Down syndrome).
* Inability or unwillingness of research participant or legal - guardian/representative to give written informed consent.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inventory of Parent and Peer Attachment (IPPA). | Baseline
  This is a self-report measure of perceptions of the relationship between an individual and their mother, father and close friends.
UCLA Loneliness Scale. | Baseline
  This 20-item self-report questionnaire assesses perceptions of peer connectedness over the past month. Items assess feelings of social connectedness, loneliness, and social isolation. Questions are answered on a 4-point Likert scale from "never" to "often," and a total score is calculated.
Family Management Measure (FMM). | Baseline
  This is a 53-item measure for parents designed to assess the impact of a child's health condition on the family system. Six subscales are derived, including measures of the child's daily life, the parent's perceived ability to manage the condition, and, for partnered parents, how the parents work together to manage the condition.
Self-Perception Profile for Adolescents/Emerging Adults (SPPA/EA). | Baseline
  The SPPA/EA is a self-report measure of self-competence. Multiple constructs are assessed, including social, romantic, physical, and academic competence, as well as global self-worth. Subscales assessing Social Competence, Romantic Competence and Physical Appearance are of primary interest.
NIH Toolbox - Friendship | Baseline
  This is a 5- (ages 15-17) or 8-item (ages 18+) self- report questionnaire that assesses aspects of friendship. Questions assess perceived ability to access friend and participation in activities with friends over the past month on a 5-point Likert scale from never to always. Five items are similar across the two age groups. Raw scores are converted to T-scores (M = 50, SD = 10), with higher scores indicative of more perceived friends to interact with.

SECONDARY OUTCOMES:
Young Adult Cancer Impact Scale | Baseline
  This is a 5-item self-report measure that assesses an individual's perception of the impact of cancer on relevant domains: education, social interaction, career goals, romantic relationships and independent living. Items are rated on a 1-10 scale from "did not interfere/affect" to "extremely interfered/affected." The social interaction and romantic relationship items are of primary interest.
Centrality of Events (COE). | Baseline
  The COE is a 20-item self-report measure that assesses an individual's perception of the impact that a traumatic or significant event as had on their identity development. Participants will be asked to complete the COE based on their experiences with cancer.
Online Social Support Scale (OSSS). | Baseline
  The two part OSSS assesses the role of online apps or websites in an individual's perception of the support they receive from others. In the first part, participants rate the frequency that they use specific online spaces (e.g., Instagram, Twitter, Facebook) to interact with others. Space is also provided for participants to free text additional sites. In the second part, 40 items assess the types of social support individuals receive from these spaces, with four subscales derived: Esteem/Emotional Support, Social Companionship, Informational Support, and Instrumental Support. Oneline Social Support Scale-scores could range from 0 to 160 with higher scores indicating receipt of more support.
Multidimensional Scale of Perceived Social Support (MSPSS). | Baseline
  The MSPSS is a 12-item self-report questionnaire that assesses perceived reception of support from important persons - friends, family, and significant other. Questions are answered on 7-item Likert scale from "very strong disagree" to "very strongly agree." Higher scores are indicative of more social support.
Responses to Stress Questionnaire (RSQ) | Baseline
  The RSQ is a 57-item self-report questionnaire assessing an individual's coping with an identified stressor. For this study, cancer will be the identified stressor and separate versions of the RSQ are available for those on treatment and off treatment. Responses to Stress Questionnaire - scores range from 0 to 4 with higher scores indicating more use of that coping mechanism
PROMIS Profile / Pediatric Profile | Baseline
  Three brief self-report measures will assess symptoms of anxiety, depression, and fatigue over the past 7 days. Measures will be completed by both AYA and their caregivers, with each respondent providing indicators of their own level of distress. Raw scores are converted to T- scores (M = 50, SD = 10) with higher scores indicating greater symptoms.
PedsQL - Cancer Specific Module | Baseline
  The PedsQL Cancer Module is a 27-item self-report measure that assesses symptom burden and quality of life as related to cancer-specific factors, including pain, nausea, procedural anxiety, and physical appearance. AYA will complete this measure as an indicator of current cancer- related symptoms. PedsQL - scores range 0 to 100 with higher scores indicating better functioning
PedsQL - Core Module | Baseline
  The PedsQL Core Module is a 23-item measure of quality of life, with both self- and proxy-report versions available. Four subscales provide two broad domains - Physical and Psychosocial Functioning - and an overall quality of life score. Raw scores undergo a linear transformation. AYA and their participating caregiver will complete this measure.
Intensity of Treatment (ITR-3). | Baseline
  The ITR-3 is a clinician-completed rating form that provides a means of classifying the intensity of pediatric cancer treatment. Four categories are elicited: Least, Moderately, Very, and Most Intensive. This will be completed for each participant using information gathered from the medical record.
Needs Assessment | Baseline
  This is a new questionnaire developed specifically for this study. Participants will answer questions about their participation in current hospital activities and events as well as their interest in and feedback on future interventions. It will be analyzed at the individual item level.
Qualitative Interview | Baseline
  A subsample of participants will complete an interview to further assess aspects of friendships and intervention interest. Participant responses will be transcribed and analyzed for themes.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah W. Daniels, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT04328350/ICF_000.pdf